CLINICAL TRIAL: NCT01922791
Title: Placebo-controlled Intervention Study for Maternal and Child Health
Brief Title: Nutrition and Pregnancy Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Principal Investigator, Kirsi Laitinen, Associate professor, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: T166/2012
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Pregnancy; Obesity; Gestational Diabetes Mellitus; Adiposity; Type2 Diabetes; Cardiovascular Risk Factor; Eating Behavior; Liver Diseases; Neurodevelopmental Disorders; Cognitive Developmental Disorders
Keywords: Nutrition; Probiotics; Fish oil
MeSH Terms: conditions — Obesity; Diabetes, Gestational; Feeding Behavior; Liver Diseases; Neurodevelopmental Disorders | interventions — Fish Oils; Lacteol; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Probiotic (Active Comparator): Comparison of probiotics, fish oil and their combination to placebo
  Interventions: Dietary Supplement: Comparison of probiotics, fish oil and their combination to placebo
- Fish oil (Active Comparator): Comparison of probiotics, fish oil and their combination to placebo
  Interventions: Dietary Supplement: Comparison of probiotics, fish oil and their combination to placebo
- Probiotics and Fish oil (Active Comparator): Comparison of probiotics, fish oil and their combination to placebo
  Interventions: Dietary Supplement: Comparison of probiotics, fish oil and their combination to placebo
- Placebo (Placebo Comparator): Comparison of probiotics, fish oil and their combination to placebo
  Interventions: Dietary Supplement: Comparison of probiotics, fish oil and their combination to placebo

INTERVENTIONS:
Dietary Supplement: Comparison of probiotics, fish oil and their combination to placebo — Double-blind randomized placebo controlled intervention
  Other Names: Lactobacillus and Bifidobacterium; Fish oil; Placebo, microcrystalline cellulose; Placebo, medium-chain triglycerides

SUMMARY:
A randomized double-blind placebo controlled intervention study with pregnant obese women (n=440) will be conducted. The intervention will involve consumption of fish oil and/or probiotic capsules from early pregnancy until 6 months after delivery.

The aim of the study is firstly to investigate the effects of the supplements on the risk of gestational diabetes mellitus and obesity in the women and secondly to modify the risk markers of allergy and obesity in children of the women. Also the underlying metabolic mechanisms will be investigated.

Follow up visits at child's age of 5 to 6 years will be conducted to evalute long-term effects on maternal and child health. The aim is to investigate the impact of dietary intervention, diet, maternal overweight/obesity and gestational diabetes status as well as gut microbiota and metabolism during pregnancy on maternal and child's health, allergy and child neuropsychological development.

ELIGIBILITY:
Inclusion Criteria:

* pregnant, less than 17 gestational weeks
* overweight
* healthy

Exclusion Criteria:

* Diabetes (type 1 or 2)
* Coeliac disease
* Increased bleeding tendency

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 439 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of gestational diabetes mellitus, GDM | Assessed at gestational weeks 24-28
Fasting glucose levels | assessed at the third trimester of pregnancy
Prevalence of allergy in child | assessed at 12 and 24 months of age

SECONDARY OUTCOMES:
Need for medication for management of gestational diabetes mellitus GDM (insulin or metformin) | During pregnancy
Body composition of mother | During and after pregnancy
Immunologic and metabolic markers | During and after pregnancy
Fecal microbiota | Before, during and after intervention
Fasting serum glucose (mmol/l) (mother/ child) | Assessed at 5-6 years postpartum
Fasting serum insulin (mU/l) (mother/child) | Assessed at 5-6 years postpartum
Number of women with prediabetes using criteria defined by American Diabetes Association | Assessed at 5-6 years postpartum
Number of women with metabolic syndrome using criteria defined by The International Diabetes Federation | Assessed at 5-6 yrs postpartum
Risk for Type 2 diabetes using questionnaire (mother) | Assessed at 5-6 yrs postpartum
Serum high sensitive C-reactive protein (mg/l) (mother/child) | Assessed at 5-6 yrs postpartum
Lipid metabolism (fasting cholesterol (mmol/l), fasting triglycerides (mmol/l), fasting HDL-cholesterol (mmol/l), fasting LDL-cholesterol (mmol/l) (mother/child) | Assessed at 5-6 yrs postpartum
Serum metabolomics by NMR (mother/child) | assessed at 5-6 yrs postpartum
Obesity by body mass index (mother/child) and body fat percentage by air displacement plethysmography (mother/child) | Assessed at 5-6 yrs postpartum
Carotid intima media thickness by ultra sound (mother/child) | Assessed at 5-6 yrs postpartum
Retinal microvasculature by digital retinal imaging (mother) | Assessed at 5-6 yrs postpartum
Liver fat by ultra sound (mother) | Assessed at 5-6 yrs postpartum
Liver health by ALAT (child/mother) | Assessed at 5-6 yrs postpartum
Fecal microbiota composition (mother/child) | Assessed at 5-6 yrs postpartum
Dietary intake of foods and nutrients and diet pattern calculated from food diaries, dietary quality index and food frequencies (assessed by questionnaires)/mother and child | Assessed at 5-6 yrs postpartum
Eating behavior by Three Factor Eating Questionnaire, Neofobia and Comprehensive Feeding Practices Questionnaire, Child Feeding Questionnaire, Child Eating Behaviour Questionnaire (child) | Assessed at 5-6 yrs postpartum
Motor development by Movement Assessment Battery for Children and by Developmental Coordination Disorder Questionnaire 2007 (DCDQ'07) (Child) | Assessed at 5-6 yrs postpartum
Cognitive development by Cantab test and Wechsler Preschool and Primary Scale of Intelligence (child) | Assessed at 5-6 yrs postpartum
Child effortful/emotionally-driven inhibition by the Forbidden Toy task and by Delay of gratification test (child) | Assessed at 5-6 yrs postpartum
Social emotional assessment by Behavior Rating Inventory of Executive Functions (child) | Assessed at 5-6 yrs postpartum
The child's social competence by Multisource Assessment of Children's Social Competence questionnaire and children's behavioral, social, and attention problems by the Child Behavior Checklist. (child) | Assessed at 5-6 yrs postpartum
Infant temperament, Child Behavior Questionnaire (child) | Assessed at 5-6 yrs postpartum
Child growth measured from weight (kg) and length (cm) | Assessed at 5-6 yrs postpartum
Atopy by serum antigens and asthma by spirometry (child) | Assessed at 5-6 yrs postpartum
Immunological cells from blood (child) | Assessed at 5-6 yrs postpartum
Physical activity by questionnaires and activity monitor | Assessed at 5-6 yrs postpartum

OTHER OUTCOMES:
Body composition, growth, development and metabolic markers of the child | 0 to 24 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi Laitinen, Principal Investigator — University of Turku
Locations (2):
- Finland (2):
  - University of Turku, Turku
  - Turku University Hospital, Turku

REFERENCES:
- [Derived] Houttu V, Mongad D, Houttu N, Saros L, Zhang C, Viitaharju J, Vahlberg T, Lahti L, Laitinen K. The Impact of Maternal Supplementation of Fish Oil and/or Probiotics During Pregnancy on the Serum Metabolomic Profile From Infancy to Childhood: Secondary Analysis of a Randomized Placebo-Controlled Trial. Curr Dev Nutr. 2025 Sep 9;9(10):107553. doi: 10.1016/j.cdnut.2025.107553. eCollection 2025 Oct. PMID 41127037
- [Derived] Muhli E, Vahlberg T, Saros L, Houttu N, Pellonpera O, Tertti K, Laitinen K. Postpartum Body Composition in Women With Overweight: Associations With Diet During Pregnancy. Obes Sci Pract. 2025 Oct 13;11(5):e70093. doi: 10.1002/osp4.70093. eCollection 2025 Oct. PMID 41098558
- [Derived] Saros L, Vahlberg T, Koivuniemi E, Houttu N, Tertti K, Shivappa N, Hebert JR, Niinikoski H, Laitinen K. Maternal diet and gestational diabetes mellitus modestly influence children's growth during their first 24 months. J Pediatr Gastroenterol Nutr. 2025 Aug;81(2):355-366. doi: 10.1002/jpn3.70098. Epub 2025 Jun 9. PMID 40491247
- [Derived] Lotankar M, Houttu N, Benchraka C, Lahti L, Laitinen K. Links between gut microbiota with specific serum metabolite groups in pregnant women with overweight or obesity. Nutr Metab Cardiovasc Dis. 2025 Sep;35(9):104095. doi: 10.1016/j.numecd.2025.104095. Epub 2025 Apr 16. PMID 40348632
- [Derived] Saros L, Setanen S, Hieta J, Kataja EL, Suorsa K, Vahlberg T, Tertti K, Niinikoski H, Stenholm S, Jartti T, Laitinen K. The effect of maternal risk factors during pregnancy on children's motor development at 5-6 years. Clin Nutr ESPEN. 2025 Apr;66:236-244. doi: 10.1016/j.clnesp.2025.01.047. Epub 2025 Jan 25. PMID 39870192
- [Derived] Saros L, Vahlberg T, Koivuniemi E, Houttu N, Niinikoski H, Tertti K, Laitinen K. Fish Oil And/Or Probiotics Intervention in Overweight/Obese Pregnant Women and Overweight Risk in 24-Month-Old Children. J Pediatr Gastroenterol Nutr. 2023 Feb 1;76(2):218-226. doi: 10.1097/MPG.0000000000003659. Epub 2022 Nov 23. PMID 36705702
- [Derived] Houttu N, Mokkala K, Saleem WT, Virtanen S, Juhila J, Koivuniemi E, Pellonpera O, Tertti K, Luokola P, Sorsa T, Salonen A, Lahti L, Laitinen K. Potential pathobionts in vaginal microbiota are affected by fish oil and/or probiotics intervention in overweight and obese pregnant women. Biomed Pharmacother. 2022 May;149:112841. doi: 10.1016/j.biopha.2022.112841. Epub 2022 Mar 28. PMID 35344737
- [Derived] Lotankar M, Mokkala K, Houttu N, Koivuniemi E, Sorensen N, Nielsen HB, Munukka E, Lahti L, Laitinen K. Distinct Diet-Microbiota-Metabolism Interactions in Overweight and Obese Pregnant Women: a Metagenomics Approach. Microbiol Spectr. 2022 Apr 27;10(2):e0089321. doi: 10.1128/spectrum.00893-21. Epub 2022 Mar 28. PMID 35343768
- [Derived] Mokkala K, Gustafsson J, Vahlberg T, Vreugdenhil ACE, Ding L, Shiri-Sverdlov R, Plat J, Laitinen K. Serum CathepsinD in pregnancy: Relation with metabolic and inflammatory markers and effects of fish oils and probiotics. Nutr Metab Cardiovasc Dis. 2022 May;32(5):1292-1300. doi: 10.1016/j.numecd.2022.02.011. Epub 2022 Feb 23. PMID 35304048
- [Derived] Pajunen L, Korkalo L, Koivuniemi E, Houttu N, Pellonpera O, Mokkala K, Shivappa N, Hebert JR, Vahlberg T, Tertti K, Laitinen K. A healthy dietary pattern with a low inflammatory potential reduces the risk of gestational diabetes mellitus. Eur J Nutr. 2022 Apr;61(3):1477-1490. doi: 10.1007/s00394-021-02749-z. Epub 2021 Nov 30. PMID 34846602
- [Derived] Davidson SJ, Barrett HL, Price SA, Callaway LK, Dekker Nitert M. Probiotics for preventing gestational diabetes. Cochrane Database Syst Rev. 2021 Apr 19;4(4):CD009951. doi: 10.1002/14651858.CD009951.pub3. PMID 33870484
- [Derived] Mokkala K, Houttu N, Koivuniemi E, Sorensen N, Nielsen HB, Laitinen K. GlycA, a novel marker for low grade inflammation, reflects gut microbiome diversity and is more accurate than high sensitive CRP in reflecting metabolomic profile. Metabolomics. 2020 Jun 20;16(7):76. doi: 10.1007/s11306-020-01695-x. PMID 32564244
- [Derived] Mokkala K, Vahlberg T, Pellonpera O, Houttu N, Koivuniemi E, Laitinen K. Distinct Metabolic Profile in Early Pregnancy of Overweight and Obese Women Developing Gestational Diabetes. J Nutr. 2020 Jan 1;150(1):31-37. doi: 10.1093/jn/nxz220. PMID 31529056
- [Derived] Pellonpera O, Mokkala K, Houttu N, Vahlberg T, Koivuniemi E, Tertti K, Ronnemaa T, Laitinen K. Efficacy of Fish Oil and/or Probiotic Intervention on the Incidence of Gestational Diabetes Mellitus in an At-Risk Group of Overweight and Obese Women: A Randomized, Placebo-Controlled, Double-Blind Clinical Trial. Diabetes Care. 2019 Jun;42(6):1009-1017. doi: 10.2337/dc18-2591. Epub 2019 Apr 9. PMID 30967436
- [Derived] Mokkala K, Roytio H, Munukka E, Pietila S, Ekblad U, Ronnemaa T, Eerola E, Laiho A, Laitinen K. Gut Microbiota Richness and Composition and Dietary Intake of Overweight Pregnant Women Are Related to Serum Zonulin Concentration, a Marker for Intestinal Permeability. J Nutr. 2016 Sep;146(9):1694-700. doi: 10.3945/jn.116.235358. Epub 2016 Jul 27. PMID 27466607
- See also: University of Turku — http://www.utu.fi
- See also: Turku University Hospital — http://www.tyks.fi
- See also: Research group www-pages — https://sites.utu.fi/nutritionresearch/